CLINICAL TRIAL: NCT05924932
Title: Effect of an Artificial Pancreas System on Glycemic Control in Patients With Type 1 Diabetes
Brief Title: Effect of HCL Insulin Delivery System on Glycemic Control in Patients With T1D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Lucie Radovnická, MD, Masaryk Hospital Usti nad Labem
Other Study IDs: Masaryk Hospital
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes mellitus; hybrid closed loop system for automatic insulin dosing; glycated hemoglobin
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for measurement of glycated hemoglobin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- group 1 with Control IQ system: Tandem t:slim X2 with hybrid closed loop system Control IQ, glucose sensor: Dexcom G6
  Interventions: Device: Tandem t:slim X2 with hybrid closed loop system Control IQ, glucose sensor: Dexcom G6
- Group 2 with SmartGuard system: MiniMed 780G, with hybrid closed loop system SmartGuard, sensor Guardien 4
  Interventions: Device: MiniMed 780G, with hybrid closed loop system SmartGuard, sensor Guardien 4

INTERVENTIONS:
Device: Tandem t:slim X2 with hybrid closed loop system Control IQ, glucose sensor: Dexcom G6 — type of hybrid close loop insulin delivery system
  Other Names: Control IQ
  Groups: group 1 with Control IQ system
Device: MiniMed 780G, with hybrid closed loop system SmartGuard, sensor Guardien 4 — type of hybrid close loop insulin delivery system
  Other Names: SmartGuard
  Groups: Group 2 with SmartGuard system

SUMMARY:
The goal of this study is compare the effect of hybrid closed loop system (HCL) for automatic insulin dosing treatment on the glycemic control of type 1 diabetes (T1D) in patient with different initial glycated hemoglobin.

DETAILED DESCRIPTION:
Rationale for the Study:

According to our hypothesis, even T1D patients with an initially optimal glucose level should benefit from this treatment method in the form of a reduction in glycemic variability.

There are very few clinical studies from real practice in a larger group of patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with T1D
* Type 1 diabetes for > 1 years
* ≥ 18 years old
* CSII (without HCL) or MDI

Exclusion Criteria:

* Severe noncompliance
* Known severe diabetic retinopathy and/or macular edema,
* Lactation, pregnancy, or intending to become pregnant during the study;
* A condition likely to require MRI. Use of acetaminophen-containing medication;
* Unwillingness to use the study device for >70% of time.
* Conditions that affect red blood cell turnover (hemolytic and other anemias, glucose-6-phosphate dehydrogenase deficiency, recent blood transfusion, use of drugs that stimulate erythropoesis, end-stage kidney disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with Type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
glycated hemoglobin | 12 month
  The difference and changes in glycated hemoglobin (HbA1c, % DCCT [mmol/mol]) between baseline and at 12 months after using HCL.

SECONDARY OUTCOMES:
tim spent in TIR | 12 month
  changes in percentage of time in range (%TIR, 70-180 mg/dL [3.9-10.0 mmol/L])
time spent in hypoglycemia | 12 month
  percentage of time spent in hypoglycemia (%TBR, <70 mg/dL [<3.9 mmol/L] and <54 mg/dL [<3.0 mmol/L])
time spent in hyperglycemia | 12 month
  percentage of time spent in hyperglycemia (%TAR, >180 mg/dL [>10.0 mmol/L] and >250 mg/dL [>13.9 mmol/L])
glycemic variability | 12 m,onth
  glycemic variability expressed as the percentage coefficient of variation (%CV) and standard deviation (SD)
mean sensor glucose value | 12 month
  mean sensor glucose value

OTHER OUTCOMES:
Safety and Tolerability | 12 month
  the incidence of severe hypoglycemia (requiring third-party assistance to treat), ketoacidosis requiring hospitalization, skin reaction, infection, or hematoma at the site of insertion of the sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Lastuvka, Study Chair — Masaryk hospital
Locations (1):
- Lucie Radovnická, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Leelarathna L, Choudhary P, Wilmot EG, Lumb A, Street T, Kar P, Ng SM. Hybrid closed-loop therapy: Where are we in 2021? Diabetes Obes Metab. 2021 Mar;23(3):655-660. doi: 10.1111/dom.14273. Epub 2020 Dec 20. PMID 33269551
- [Result] Bergenstal RM, Nimri R, Beck RW, Criego A, Laffel L, Schatz D, Battelino T, Danne T, Weinzimer SA, Sibayan J, Johnson ML, Bailey RJ, Calhoun P, Carlson A, Isganaitis E, Bello R, Albanese-O'Neill A, Dovc K, Biester T, Weyman K, Hood K, Phillip M; FLAIR Study Group. A comparison of two hybrid closed-loop systems in adolescents and young adults with type 1 diabetes (FLAIR): a multicentre, randomised, crossover trial. Lancet. 2021 Jan 16;397(10270):208-219. doi: 10.1016/S0140-6736(20)32514-9. PMID 33453783